CLINICAL TRIAL: NCT00768885
Title: Comparative Study of the Wearing Satisfaction of Two Soft Contact Lens Designs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: MDPTLD0809
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PureVision 1 (Active Comparator): PureVision soft contact lens design #1.
  Interventions: Device: PureVision 1
- PureVision 2 (Experimental): PureVision soft contact lens design #2
  Interventions: Device: PureVision 2

INTERVENTIONS:
Device: PureVision 1 — Currently marketed PureVision soft contact lens.
  Arms: PureVision 1
Device: PureVision 2 — Alternate design soft contact lens.
  Arms: PureVision 2

SUMMARY:
To evaluate the wearing satisfaction of a new design of the PureVision soft contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Subject is myopic
* Subjects who wear soft contact lenses that are exchanged at least biweekly at the time consent is obtained.

Exclusion Criteria:

* Systemic disease affecting ocular health
* Using pharmaceuticals that may affect the function of the eyes or lenses.
* Subject possessing corneal infiltrate or corneal ulcers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kodama Eye Clinic, Kyoto, Japan